CLINICAL TRIAL: NCT04082091
Title: Screening, Early Referral and Lifestyle Tailored E_prescription for Cardiovascular Prevention in PakisTan(SELECT) - A Pilot Feasibility Study Using mHealth
Brief Title: Screening, Early Referral and Lifestyle Tailored E_prescription for Cardiovascular Prevention
Acronym: SELECT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Collaborators: The George Institute (Other)
Responsible Party: Principal Investigator, Dr. Ayeesha Kamran Kamal, Professor of Neurology, Department of Medicine, Aga Khan University
Other Study IDs: 2019-0599-2619
Record Dates: First submitted 2019-09-03; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Cardiovascular Diseases; Cerebral Infarction; Type2 Diabetes Mellitus; Hypertension,Essential; Prevention
Keywords: mHealth; mixed method; feasibility study; Malir district
MeSH Terms: conditions — Cardiovascular Diseases; Cerebral Infarction; Essential Hypertension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: SELECT mHealth Program — Individuals will be screened via the telephone, using a mobile-based algorithm that prompts questions about hypertension, risk of Diabetes Mellitus, use of smokeless tobacco and smoking, level of physical activity, and main nutritional choices. These questions are based on tools that have been validated in studies undertaken in this population and will be directly administered by trained research staff of Aga Khan University. Screening will prompt triage into three categories: "high" - referred to the conveniently located integrated medical center for a medical teleconsultation and fasting glucose test; "medium" - receive fasting glucose test and BP measurement; and "low" risk. All subjects in each category will be enrolled in an e_Prescription intervention for lifestyle change tailored to their individual risk profile.

SUMMARY:
We will evaluate an e_Prescription intervention can be integrated into an electronic screening program, which together exploit: (i) reach - the adult population has 100% mobile phone ownership and 92% internet national coverage; and (ii) behavioral change - the intervention can teach verbally and visually, thus bypassing literacy challenges, to allow simple, low-cost, repetition messaging for habit reinforcement. Uptake of the program through the various stages will be evaluated in ~2000 adults of a large representative suburban district of Karachi: As well as before-and-after physiological measures, including blood pressure (BP) and blood glucose, a random sample of 30-40 participants will be invited for interview to assess success and failure of the program. This is a pragmatic feasibility intervention implementation study.

DETAILED DESCRIPTION:
The goal of this pilot study is to demonstrate feasibility of a scalable , population-wide, approach to early detection and management of people at high-risk of CVD using electronic screening, referral, treatment and lifestyle modification based on health theory and considerable background research for local applicability.

It is a mixed method, feasibility study based in Malir District of Karachi, the largest city in Pakistan, to demonstrate uptake, participation and response of our mHealth intervention.

ELIGIBILITY:
Inclusion Criteria:

* All adult (>18 years) residents of Malir district
* Own a mobile phone
* Provide written informed consent are eligible to participate

Exclusion Criteria:

* Not permanent residents of Malir district.
* A person who is decision impaired due to stroke, or aphasia or dementia .
* Serious cognitive deficits that impair the visualization or understanding of SMS, IVR and e_prescription messages

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The pilot study will be undertaken in the Malir area (80,000 persons), one of the largest districts of Karachi (population 120 million), with urban, urban slum, and rural urban areas, and includes all ethnicities and economic strata of Pakistan. In this location, the Aga Khan University Health System, one of the major health systems of Pakistan, has integrated medical centers (IMSs) with laboratory testing, resident physicians, and ability to triage and refer people to a main tertiary hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Health Service Delivery of Intervention Outreach via Short Text Messages | 3 to 6 months
  The success rate in delivery of SMS intervention to target community
  1. Number of SMS sent successfully to target Population
Health Service Delivery of Intervention Outreach via Interactive Voice Recording | 3 to 6 months
  Number of IVR ( Interactive Voice Recording ) sent to target Population
Health Service Measures of Intervention Uptake | 3 to 6 months
  Proportion of referred participants enrolled in e_Prescription education program
Community Participation and Uptake of Intervention | 3 to 6 months
  Number of participants responded to the IVR and SMS call
Early Impact Measure of Intervention for Prompt Referral | 3 to 6 months
  Proportion of referred participants from screened participants referred
Early Impact Measure of Intervention for Detection | 3 to 6 months
  Proportion of participants in each of risk strata (low, medium and high risk) as defined by
  the presence of stroke and/or MI ( High ), DM and / or HTN ( Medium), or poor lifestyle choices ( Low Risk) by the SELECT algorithm

SECONDARY OUTCOMES:
Change in Physiological Characteristics of Intervention Participants - Blood Pressure | 0, 3 to 6 months
  Mean difference in systolic and diastolic Blood Pressure before and after intervention in mm Hg.
Change in Physiological Characteristics of Intervention Participants - Weight | 0, 3 to 6 months
  Mean difference in weight before and after intervention in kg
Change in Physiologic Characteristics of Intervention Participants- Height | 0, 3 to 6 months
  Height in metres to determine Body Mass Index ( BMI )
Change in Physiological Characteristics of Intervention Participants - BMI | 0, 3 to 6 months
  Mean difference in BMI before and after intervention in kg/m2
Change in Physiological Characteristics of Intervention Participants - Physical Activity | 0, 3 to 6 months
  Increase in number of hours in physical activity from baseline (self-reported) measured by the IPAQ Short scale self reported version ( International Physical Activity Questionnaire) which will report low medium and high levels of physical activity based on 600 MET minutes /week ( Moderate),1500- 3000 MET minutes /week ( High), and low as any value less than the above.

CONTACTS AND LOCATIONS:
Overall Officials: Ayeesha Kamal, MD, Principal Investigator — Aga Khan University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jafar TH, Haaland BA, Rahman A, Razzak JA, Bilger M, Naghavi M, Mokdad AH, Hyder AA. Non-communicable diseases and injuries in Pakistan: strategic priorities. Lancet. 2013 Jun 29;381(9885):2281-90. doi: 10.1016/S0140-6736(13)60646-7. Epub 2013 May 17. PMID 23684257
- [Background] Kamal AK, Khoja A, Usmani B, Muqeet A, Zaidi F, Ahmed M, Shakeel S, Soomro N, Gowani A, Asad N, Ahmed A, Sayani S, Azam I, Saleem S. Translating knowledge for action against stroke--using 5-minute videos for stroke survivors and caregivers to improve post-stroke outcomes: study protocol for a randomized controlled trial (Movies4Stroke). Trials. 2016 Jan 27;17:52. doi: 10.1186/s13063-016-1175-x. PMID 26818913
- [Background] Mohan V, Deepa R, Deepa M, Somannavar S, Datta M. A simplified Indian Diabetes Risk Score for screening for undiagnosed diabetic subjects. J Assoc Physicians India. 2005 Sep;53:759-63. PMID 16334618
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Khan M, Kamal AK, Islam M, Azam I, Virk A, Nasir A, Rehman H, Arif A, Jan M, Akhtar A, Mawani M, Razzak JA, Pasha O. Can trained field community workers identify stroke using a stroke symptom questionnaire as well as neurologists? Adaptation and validation of a community worker administered stroke symptom questionnaire in a peri-urban Pakistani community. J Stroke Cerebrovasc Dis. 2015 Jan;24(1):91-9. doi: 10.1016/j.jstrokecerebrovasdis.2014.07.030. Epub 2014 Oct 16. PMID 25440346
- [Background] Rahman MA, Spurrier N, Mahmood MA, Rahman M, Choudhury SR, Leeder S. Rose Angina Questionnaire: validation with cardiologists' diagnoses to detect coronary heart disease in Bangladesh. Indian Heart J. 2013 Jan-Feb;65(1):30-9. doi: 10.1016/j.ihj.2012.09.008. Epub 2012 Sep 12. PMID 23438610